CLINICAL TRIAL: NCT05205811
Title: A Randomized Controlled Trial to Determine the Effects of Combination Zonisamide and Bupropion on Switching to an Electronic Cigarette
Brief Title: The Effects of Combination Zonisamide and Bupropion on Switching to an Electronic Cigarette
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BuZonE 2
Record Dates: First submitted 2021-10-27; First posted 2022-01-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Smoking Cessation
Keywords: e-cigarette; zonisamide; bupropion; combustible cigarettes
MeSH Terms: conditions — Smoking Cessation; Vaping | interventions — Bupropion; Zonisamide; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Combination zonisamide and bupropion with e-cigarette (Experimental): After the first week of e-cigarette use (JUUL), participants will be given bupropion (150 mg each morning for days 1-3, then 300 mg daily) with zonisamide (100 mg daily). The combination of zonisamide and bupropion use will continue for 7 weeks of treatment, and e-cigarette use will continue until the end of the study (an additional 4 weeks).
  Interventions: Drug: Bupropion; Drug: Zonisamide; Other: E-cigarette
- Bupropion with e-cigarette (Experimental): After the first week of e-cigarette use (JUUL), participants will be given bupropion (150 mg each morning for days 1-3, then 300 mg daily) with placebo zonisamide. The combination of placebo and bupropion use will continue for 7 weeks of treatment, and e-cigarette use will continue until the end of the study (an additional 4 weeks).
  Interventions: Drug: Bupropion; Drug: Placebo zonisamide; Other: E-cigarette
- Placebo with e-cigarette (Placebo Comparator): After the first week of e-cigarette use (JUUL), participants will be given placebo bupropion with placebo zonisamide. The combination of these placebos will continue for 7 weeks of treatment, and e-cigarette use will continue until the end of the study (an additional 4 weeks).
  Interventions: Drug: Placebo bupropion; Drug: Placebo zonisamide; Other: E-cigarette

INTERVENTIONS:
Drug: Bupropion — Extended-release bupropion dosing (150 mg each morning days 1-3, then 300 mg/daily) for the remainder of the 7 weeks.
  Other Names: Wellbutrin; Zyban
  Arms: Bupropion with e-cigarette; Combination zonisamide and bupropion with e-cigarette
Drug: Zonisamide — Zonisamide (100 mg/daily) for 7 weeks.
  Other Names: zonegran
  Arms: Combination zonisamide and bupropion with e-cigarette
Drug: Placebo bupropion — Placebo bupropion for 7 weeks.
  Arms: Placebo with e-cigarette
Drug: Placebo zonisamide — Placebo zonisamide for 7 weeks.
  Arms: Bupropion with e-cigarette; Placebo with e-cigarette
Other: E-cigarette — e-cigarette for ad libitum use for two weeks prior to complete switch day and for an additional 10 weeks.
  Other Names: JUUL

SUMMARY:
This three-group randomized double-blind placebo-controlled trial (N=180) will evaluate the impact of combination zonisamide and bupropion on the process of switching from combustible cigarettes (CCs) to an e-cigarette. There will be a data collection period of at least five days to obtain baseline information on the use of combustible cigarettes. All participants enrolled in the study will receive a JUUL e-cigarette at Visit 2 for ad libitum use. After the first week of e-cigarette use (at Visit 3), participants will be given bupropion (150 mg each morning for days 1-3, then 300 mg daily) with either zonisamide (100 mg daily) or placebo (group 1 and group 2 respectively), or placebo for both medications (group 3) in addition to continued use of the e-cigarette. At each visit, participants will receive enough study drugs (or placebos) and e-cigarettes to last until their next study visit. The combination of zonisamide and bupropion use will continue until Visit 6 (7 weeks of treatment), and e-cigarette use will continue until the end of treatment (Visit 7).

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the ICF and is able to read and understand the information provided in the ICF.
2. Is 21 to 65 years of age (inclusive) at screening.
3. Smokes at least 10 commercially available cigarettes per day (no brand restrictions), for the last 12 months.
4. Has an expired air CO reading of at least 10 ppm at screening.
5. Is interested in switching to an electronic cigarette.
6. Is willing and able to comply with the requirements of the study.
7. Owns a smartphone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., safety laboratory, vital signs, physical examination, ECG, concomitant medications and medical history).
2. Has a PHQ-9 score greater than 9, or a score greater than 0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") at screening.
3. Has plans to use an FDA-approved smoking cessation product during the study.
4. Has high blood pressure (systolic > 150 mmHg or diastolic >95 mmHg) at screening.
5. Has body mass index (BMI) less than 15.0 kg/m2 or greater than 40.0 kg/m2.
6. Has coronary heart disease, structural cardiac disease (including, but not limited to valvular heart disease or cardiac murmurs), cardiac dysrhythmias, syncope, cardiac chest pain, or history of heart attack or heart failure.
7. Has received psychotherapy or behavioral treatments potentially impacting symptoms of depression, anxiety, or nicotine withdrawal within 30 days of screening, or during the study.
8. Is taking antidepressants, psychoactive medications (e.g. antipsychotics, benzodiazepines, hypnotics) or medications that prolong QTc.
9. Has used any of these products in the past 30 days:

   1. Illegal drugs (or if the urine drug screen is positive for cocaine, THC, amphetamines, methamphetamines, or opiates);
   2. Experimental (investigational) drugs that are unknown to participant;
   3. Chronic opiate use.
10. Has used smokeless tobacco (chewing tobacco, snuff), cigars (except for "Black & Mild" cigars or Cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of screening.
11. Has a plan to use an FDA-approved quit-smoking treatment in the next 30 days.
12. Is pregnant or nursing (by self-report) or has a positive pregnancy test.
13. Enrollment requirements met.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Complete Switching From Combustible Cigarettes to JUUL e-cigarette as measured by Exhaled carbon monoxide (CO) | After 8 weeks
  Exhaled carbon monoxide (CO) < 5 ppm at the end of drug treatment
Complete Switching From Combustible Cigarettes to JUUL e-cigarette as measured by change in Total urinary 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) | Baseline, Week 8, Week 12
  Total urinary 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL)
Complete Switching From Combustible Cigarettes to JUUL e-cigarette as measured by change in self-report of daily cigarette and e-cigarette use | Daily from Week 2 to Week 12
  Self-report of daily cigarette and e-cigarette use

SECONDARY OUTCOMES:
Change in Smoking withdrawal symptoms | Baseline, Week 1, Week 2, Week 4, Week 8, Week 12
  Smoking withdrawal symptoms will be collected using a questionnaire developed by Drs. Shiffman and Jarvik (1976), which assesses craving for cigarettes, negative mood, arousal, missing the habit of smoking, changes in appetite and somatic symptoms and a seven-point scale (from 1-Not at All to 7-Extremely). Higher scores indicate more withdrawal symptoms.
Change in Rewarding and aversive effects of smoking and e-cigarette use | Baseline, Week 1, Week 2, Week 4, Week 8, Week 12
  The mCEQ-E will be utilized to assess the degree to which participants experience the reinforcing of smoking, providing five subscale scores: smoking satisfaction (satisfying, tastes good,enjoy smoking), psychological rewards (calms down, more awake, less irritable, helps concentrate, reduces hunger), aversion (dizziness, nauseated), enjoyment of respiratory tract sensations (single-item assessment), craving reduction (single-item assessment). Participants will be asked to assess the 12 items of the questionnaire on a 7-point scale, ranging from "not at all" to "extremely". These 12 items will be asked for the "first cigarette smoked", "cigarette immediately after a meal", and "all other cigarettes." The e-cigarette version of this questionnaire (mECEQ-E) will also be used.

OTHER OUTCOMES:
Tolerability of study drugs as measured by frequency of drug termination or drug non-adherence | Baseline, Week 1, Week 2, Week 4, Week 8
  The frequency of drug termination or non-adherence prior to Week 8 will be tabulated for each condition. Adverse effects will also be tabulated for each condition, including the following adverse effects of special interest (AESIs): insomnia, agitation, dry mouth, somnolence, headache, nausea, constipation, diarrhea, dizziness or loss of appetite.
Seven-day point abstinence at 6 months post-switch | 6 Months post Switch Day
  Seven-day point abstinence at 6 months post-switch will be assessed by self-report and confirmed by exhaled carbon monoxide (CO) < 5 ppm.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961